CLINICAL TRIAL: NCT00875563
Title: Evaluation of the Safety and Effectiveness of the Zenith(R) Fenestrated AAA Endovascular Graft
Brief Title: Zenith(R) Fenestrated Abdominal Aortic Aneurysm (AAA) Endovascular Graft Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 04-541; 370015, FNCT
Expanded Access: NCT02577562 (Approved for marketing)
Record Dates: First submitted 2009-02-19; First posted 2009-04-03 (Estimated); Results first posted 2015-09-30 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-03

CONDITIONS: Abdominal Aortic Aneurysms; Aorto-iliac Aneurysms; Juxtarenal Aneurysms
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

ARMS (1):
- 1 (Experimental): Zenith(R) Fenestrated AAA Endovascular Graft
  Interventions: Device: Zenith(R) Fenestrated AAA Endovascular Graft

INTERVENTIONS:
Device: Zenith(R) Fenestrated AAA Endovascular Graft — The Zenith(R) Fenestrated AAA Endovascular Graft with the H&L-B One-Shot™ Introduction System is indicated for the endovascular treatment of patients with abdominal aortic or aortoiliac aneurysms having morphology suitable for endovascular repair

SUMMARY:
The Zenith(R) Fenestrated AAA Endovascular Graft Clinical Study is a clinical investigation approved by the US FDA to study the safety and effectiveness of the Zenith(R) Fenestrated AAA Endovascular Graft in the treatment of abdominal aortic and aorto-iliac aneurysms.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal aortic and aortoiliac aneurysms with diameter greater than or equal to 5 cm

Exclusion Criteria:

* Proximal neck less than 4 mm or greater than or equal to 15 mm in length unless otherwise compromised to preclude seal
* Renal artery stenosis greater than 50 percent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2005-01; Primary Completion 2011-02 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - University of California, San Francisco, San Francisco, California
  - Shands Hospital, Gainesville, Florida
  - The Indiana Heart Hospital, Indianapolis, Indiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Massachusetts, Worcester, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - NYU Medical Center, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Harborview Medical Center, Seattle, Washington

REFERENCES:
- See also: Zenith abdominal aortic aneurysm endovascular graft — http://www.ncbi.nlm.nih.gov/pubmed/18486418

RESULTS

PARTICIPANT FLOW:
Groups:
- Zenith® Fenestrated AAA Endovascular Graft: The Zenith® Fenestrated AAA Endovascular Graft with the H&L-B One-Shot™ Introduction System is indicated for the endovascular treatment of patients with abdominal aortic or aortoiliac aneurysms having morphology suitable for endovascular repair
Period: Overall Study
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Started | 42
Completed | 18
Not Completed | 24
Not completed — Death | 4
Not completed — Withdrawal by Subject | 7
Not completed — No long-term (3-5 year) consent | 6
Not completed — Still be eligible for follow-up | 7

BASELINE CHARACTERISTICS:
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 75.3 (7.4)
Gender [Count of Participants; unit: Participants]
  Female | 9
  Male | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Success
Description: Technical success (successful access, deployment, and patency of the Fenestrated Graft, and patency of all vessels targeted by a fenestration intra-operatively), and freedom from the following: type I or type III endoleaks, AAA-related serious adverse events, AAA-related major complications, and aneurysm enlargement greater than 0.5 cm.
  A serious adverse event is defined as any occurrence of death, aneurysm rupture, or conversion to open surgical repair.
  A major complication is defined as any occurrence of Q-wave myocardial infarction, congestive heart failure, cardiac ischemia requiring intervention, renal failure requiring permanent dialysis, bowel obstruction, ischemia, or fistula, stroke with permanent deficit, or paralysis.
Time Frame: 6 months
Population: Two patients were lost to follow-up and did not have CT data at 6 months. Patients treated with the Zenith® Fenestrated AAA Endovascular Graft was compared to propensity score matched patients treated with the Zenith® AAA Endovascular Graft (NCT00196092, link to 5-year study results provided).
Measure: Number; unit: participants
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Number analyzed (Participants) | 40
participants | 39
Statistical Analysis 1: Comparison: Zenith® Fenestrated AAA Endovascular Graft; Patients treated with the Zenith® Fenestrated AAA Endovascular Graft were compared with matched patients treated with the Zenith® AAA Endovascular Graft; Test type: Non-Inferiority or Equivalence — An exact test method (Sidik K. 2003, Statistics in Medicine 22: 265-278) for matched controls was used, at a type I error rate of 0.05 and a non-inferiority margin of 10%. 38 pairs of patients were determined necessary, and the power was calculated to be 0.92; p = 0.02, Exact test for matched pairs

ADVERSE EVENTS:
Time Frame: 5 years
Arm/Group | Zenith® Fenestrated AAA Endovascular Graft
Serious Adverse Events (participants affected / at risk) | 4/42
Other Adverse Events (participants affected / at risk) | 24/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Fenestrated AAA Endovascular Graft (N=42)
Death (General disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Zenith® Fenestrated AAA Endovascular Graft (N=42)
Arrhythmia requiring intervention or new treatment (Cardiac disorders) | 6 (6)
Congestive heart failure (Cardiac disorders) | 4 (4)
Pneumonia requiring antibiotics (Respiratory, thoracic and mediastinal disorders) | 6 (8)
Creatinine rise > 2 mg/dl and > 30% from baseline on two or more follow-up tests (Renal and urinary disorders) | 5 (5)
Occlusion of a fenestrated renal vessel (Renal and urinary disorders) | 3 (3)
Renal infarct (Renal and urinary disorders) | 5 (5)
Post-procedure transfusion (Vascular disorders) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days